CLINICAL TRIAL: NCT00897078
Title: Health Effects After Leukemia (HEAL) Research Study
Brief Title: Study of Metabolic Syndrome in Young Patients Who Are Acute Lymphoblastic Leukemia Survivors and Their Healthy Siblings
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jill Simmons, Assistant Professor of Pediatrics, Vanderbilt University
Other Study IDs: CDR0000635797; VU-VICC-PED-0888; 081208
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia
Keywords: cancer survivor; healthy, no evidence of disease; long-term effects secondary to cancer therapy in children; childhood acute lymphoblastic leukemia in remission
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Banked DNA
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: laboratory biomarker analysis
  Other Names: none noted
Other: medical chart review
  Other Names: none noted
Other: metabolic assessment
  Other Names: none noted
Other: questionnaire administration — will be obtained at a single clinic visit
  Other Names: none noted
Procedure: assessment of therapy complications
  Other Names: none noted

SUMMARY:
RATIONALE: Gathering information about metabolic syndrome from young patients who have survived acute lymphoblastic leukemia (ALL) may help doctors learn more about the disease.

PURPOSE: This phase I trial is studying the metabolic syndrome in young patients who have survived acute lymphoblastic leukemia and in healthy sibling volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the prevalence of the metabolic syndrome (MS) and its component traits (i.e., obesity, hypertension, dyslipidemia, and insulin resistance) in survivors of childhood acute lymphoblastic leukemia and in healthy sibling volunteers.
* Identify host- and treatment-related risk factors for MS.

OUTLINE: This is a multicenter study.

Patients' medical charts are reviewed and patients undergo anthropometric measuring (height and weight for BMI calculation and waist and hip circumferences) and blood pressure testing. Patients also complete questionnaires on their physical activity, diet, and family history over 30-45 minutes. Blood is collected to measure cytokines (e.g., adiponectin, leptin, interleukin-6, and C-reactive protein), fasting glucose, and fasting insulin.

Healthy volunteers undergo anthropometric measuring and blood pressure testing (if they are seen in the clinic). They also complete a baseline medical history and questionnaires on their physical activity and diet.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Meets one of the following eligibility criteria:

  * Childhood acute lymphoblastic leukemia survivor

    * Less than 22 years old at diagnosis
    * Treated from 1990-2007 at one of the following locations:

      * Fred Hutchinson Cancer Research Center and/or Children's Hospital and Regional Medical Center in Seattle, WA
      * Vanderbilt Children's Hospital in Nashville, TN
    * Meets 1 of the following treatment criteria:

      * Completed conventional therapy ≥ 11 months ago and in first complete remission
      * Received an allogeneic hematopoietic cell transplantation ≥ 11 months ago and in complete remission
    * No evidence of recurrent disease
  * Healthy volunteer

    * Full sibling of enrolled cancer survivor
    * Age 8-21 (if more than 1 eligible sibling, sibling of closest age is preferred)
    * No history of cancer

PATIENT CHARACTERISTICS:

* Able to speak, read, and write English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No active treatment for graft-vs-host disease

Exclusion Criteria:

* Lack of ability to speak, read, and write English
* Active treatment for graft versus host disease

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A minimum target accrual at each institution is 25 subjects for each treatment modality and 25 siblings, for a total of 75 study participants at VCH. An attempt will be made to approach equal numbers of male and female survivors.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of the metabolic syndrome (MS) and its component traits in these patients and in healthy volunteers | 2009-2011
Host- and treatment-related risk factors for MS | 2009-2011

CONTACTS AND LOCATIONS:
Overall Officials: Jill Simmons, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee